CLINICAL TRIAL: NCT01068730
Title: Bioequivalence Study of 500 mg and 1000 mg Glucophage (Metformin) Tablets Manufactured by Bristol-Myers Squibb Relative to 500 mg and 1000 mg Diabex (Metformin) Tablets Marketed in Australia by Alphapharm Administered to Healthy Subjects in the Fed State
Brief Title: Bioequivalence Study of 500 mg and 1000 mg Glucophage (Metformin) Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CV181-120
Record Dates: First submitted 2010-02-12; First posted 2010-02-15 (Estimated); Results first posted 2012-03-29 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A (Other): 500 mg metformin (Diabex): Single oral dose of 500 mg metformin (Diabex) tablet administered in the fed condition
  Interventions: Drug: metformin (Diabex)
- Treatment B (Other): 500 mg metformin (Glucophage™): Single oral dose of 500 mg metformin (Glucophage™) tablet administered in the fed condition
  Interventions: Drug: metformin (Glucophage™)
- Treatment C (Other): 1000 mg metformin (Diabex): Single oral dose of 1000 mg metformin (Diabex) tablet administered in the fed condition
  Interventions: Drug: metformin (Diabex)
- Treatment D (Other): 1000 mg metformin (Glucophage™): A Single oral dose of 1000 mg metformin (Glucophage™) tablet administered in the fed condition
  Interventions: Drug: metformin (Glucophage™)

INTERVENTIONS:
Drug: metformin (Diabex) — Tablets, Oral, 500 mg, Once daily, single dose
  Other Names: Diabex
  Arms: Treatment A
Drug: metformin (Glucophage™) — Tablets, Oral, 500 mg, Once Daily, single dose
  Other Names: Glucophage™
  Arms: Treatment B
Drug: metformin (Glucophage™) — Tablets, Oral, 1000 mg, Once daily, single dose
  Other Names: Glucophage™
  Arms: Treatment D
Drug: metformin (Diabex) — Tablets, Oral, 1000 mg, Once daily, single dose
  Other Names: Diabex
  Arms: Treatment C

SUMMARY:
To demonstrate the bioequivalence of 500 mg and 1000 mg Glucophage tablets manufactured by BMS relative to the respective strengths of 500 mg and 1000 mg Diabex tablets marketed in Australia by Alphapharm in the fed state

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18 to 55 inclusive
* Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination, electrocardiograms (ECGs), and clinical laboratory determinations
* Body Mass Index (BMI) of 18 to 32 kg/m², inclusive. BMI = weight (kg)/ [height (m)]²

Exclusion Criteria:

* Any significant acute or chronic medical illness
* Current or recent (within 3 months) gastrointestinal disease
* Any major surgery within 4 weeks of study drug administration
* History of allergy or intolerance to metformin or other similar acting agents
* Prior exposure to metformin within 3 months of study drug administration
* Estimated creatinine clearance (Clcr) of < 80ml/min using the Cockcroft Gault formula

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2010-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PPD Development, LP, Austin, Texas, United States

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 28 participants who met all of the inclusion and none of the exclusion criteria were planned and enrolled in the study from a single site in the United States.
Pre-assignment Details: Participants were screened for eligibility within 21 days before Day 1 of period 1. On Day -1 of each period, the participants were admitted to the clinical facility and confined for 4 days. All the 28 participants were randomly assigned to 1 of 4 treatment sequences (ADBC, BACD, CBDA, or DCAB). The washout between each dose was at least 7 days.
Groups:
- Treatment Sequence ADBC: Treatment A (period 1): single oral 500-mg Diabex (metformin) tablet administered under fed condition. Treatment D (period 2): single oral 1000-mg Glucophage (metformin) tablet administered under fed condition. Treatment B (period 3): single oral 500-mg Glucophage tablet administered under fed condition. Treatment C (period 4): single oral 1000-mg Diabex tablet administered under fed condition.
- Treatment Sequence BACD: Treatment B (period 1): single oral 500-mg Glucophage tablet administered under fed condition. Treatment A (period 2): single oral 500-mg Diabex tablet administered under fed condition. Treatment C (period 3): single oral 1000-mg Diabex tablet administered under fed condition. Treatment D (period 4): single oral 1000-mg Glucophage tablet administered under fed condition.
- Treatment Sequence CBDA: Treatment C (period 1): single oral 1000-mg Diabex tablet administered under fed condition. Treatment B (period 2): single oral 500-mg Glucophage tablet administered under fed condition. Treatment D (period 3): single oral 1000-mg Glucophage tablet administered under fed condition. Treatment A (period 4): single oral 500-mg Diabex tablet administered under fed condition.
- Treatment Sequence DCAB: Treatment D (period 1): single oral 1000-mg Glucophage tablet administered under fed condition. Treatment C (period 2): single oral 1000-mg Diabex tablet administered under fed condition. Treatment A (period 3): single oral 500-mg Diabex tablet administered under fed condition. Treatment B (period 4): single oral 500-mg Glucophage tablet administered under fed condition.
Period: Period 1
Arm/Group | Treatment Sequence ADBC | Treatment Sequence BACD | Treatment Sequence CBDA | Treatment Sequence DCAB
Started | 7 | 7 | 7 | 7
Completed | 7 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Treatment Sequence ADBC | Treatment Sequence BACD | Treatment Sequence CBDA | Treatment Sequence DCAB
Started | 7 | 7 | 7 | 7
Completed | 7 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Treatment Sequence ADBC | Treatment Sequence BACD | Treatment Sequence CBDA | Treatment Sequence DCAB
Started | 7 | 7 | 7 | 7
Completed | 6 | 7 | 7 | 7
Not Completed | 1 | 0 | 0 | 0
Not completed — Personal reason | 1 | 0 | 0 | 0
Period: Period 4
Arm/Group | Treatment Sequence ADBC | Treatment Sequence BACD | Treatment Sequence CBDA | Treatment Sequence DCAB
Started | 6 | 7 | 7 | 7
Completed | 6 | 6 | 7 | 7
Not Completed | 0 | 1 | 0 | 0
Not completed — Family emergency | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Enrolled and Treated Participants: Participants who were randomly assigned to 1 of 4 treatment sequences (ADBC, BACD, CBDA, or DCAB). Treatment A: single oral 500-mg Diabex (metformin) tablet administered under fed condition. Treatment B: single oral 500-mg Glucophage tablet administered under fed condition. Treatment C: single oral 1000-mg Diabex tablet administered under fed condition.Treatment D: single oral 1000-mg Glucophage (metformin) tablet administered under fed condition.
Arm/Group | All Enrolled and Treated Participants
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.6 (11.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 16
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 24
  Black or African American | 4
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 18
Height [Mean (Standard Deviation); unit: Centimeter] | 169.54 (11.44)
Weight [Mean (Standard Deviation); unit: kg] | 77.02 (15.88)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.58 (3.64)

OUTCOME MEASURES:

1. Primary Outcome: Metformin Pharmacokinetic (PK) Parameter Area Under the Plasma Concentration Versus Time Curve From Time 0 Extrapolated to Infinity (AUC[0-inf])
Description: PK is the process by which a drug is absorbed, distributed, metabolized, and eliminated by the body. AUC (0-inf) is the area under the plasma concentration-time curve from time zero extrapolated to infinite time.
Time Frame: Periods 1, 2, 3, & 4: pre-dosing, 15, 30, 45 mins & 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36 & 48 hrs post-dosing
Population: All treated participants with evaluable PK analyses. In treatment D, AUC (0-inf) was not analysed for 1 participant who did not have a clear terminal elimination phase.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Treatment A - 500 mg Diabex: 500 mg metformin (Diabex): Single Oral dose of 500 mg Diabex tablet administered in the fed condition
- Treatment B - 500 mg Glucophage: 500 mg metformin (Glucophage™): Single Oral dose of 500 mg Glucophage tablet administered in the fed condition
- Treatment C - 1000 mg Diabex: 1000 mg metformin (Diabex): Single Oral dose of 1000 mg Diabex tablet administered in the fed condition
- Treatment D - 1000 mg Glucophage: 1000 mg metformin (Glucophage™): Single Oral dose of 1000 mg Glucophage tablet administered in the fed condition
Arm/Group | Treatment A - 500 mg Diabex | Treatment B - 500 mg Glucophage | Treatment C - 1000 mg Diabex | Treatment D - 1000 mg Glucophage
Number analyzed (Participants) | 28 | 27 | 27 | 25
ng*hr/mL | 7062.76 (26.91) | 7187.14 (25.95) | 11577.85 (27.36) | 11424.73 (29.06)
Statistical Analysis 1: Comparison: Treatment A - 500 mg Diabex vs Treatment B - 500 mg Glucophage; If there was no difference between the bioavailabilities of metformin from the 500-mg or 1000-mg Glucophage tablets manufactured by BMS and 500-mg or 1000-mg Diabex tablets manufactured in Australia by Alphapharm, then 20 subjects would have provided 99% power to conclude bioequivalence (BE) with respect to Cmax and AUC0-inf. If there was a 5% difference, then 20 subjects would have provided 97% and 99% power to conclude BE with respect to Cmax and AUC0-inf, respectively; Test type: Non-Inferiority or Equivalence — Bioequivalence was concluded if the 90% confidence intervals (CIs) for the test-to-reference ratios (B/A) and (D/C) of geometric means were entirely contained within 80% to 125% for both Cmax and AUC0-inf; Ratio (%) of Geometric LS Means = 102.58, 95% CI 2-sided [99.07 to 106.23] — Ratio=Treatment B/Treatment A. Geometric least squares (LS) means values are presented in other statistical analysis entries
Statistical Analysis 2: Comparison: Treatment C - 1000 mg Diabex vs Treatment D - 1000 mg Glucophage; If there was no difference between the bioavailabilities of metformin from the 500-mg or 1000-mg Glucophage tablets manufactured by BMS and 500-mg or 1000-mg Diabex tablets manufactured in Australia by Alphapharm, then 20 subjects would have provided 99% power to conclude BE with respect to Cmax and AUC0-inf. If there was a 5% difference, then 20 subjects would have provided 97% and 99% power to conclude BE with respect to Cmax and AUC0-inf, respectively; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio (%) of Geometric LS Means = 99.67, 95% CI 2-sided [96.16 to 103.31] — Ratio=Treatment D/Treatment C. Geometric LS means values are presented in other statistical analysis entries
Statistical Analysis 3: Comparison: Treatment A - 500 mg Diabex; Geometric least squares means for Treatment A; Test type: Superiority or Other; Geometric Least Squares Mean (ng*hr/mL) = 7062.8
Statistical Analysis 4: Comparison: Treatment B - 500 mg Glucophage; Geometric least squares means for Treatment B; Test type: Superiority or Other; Geometric Least Squares Mean (ng*hr/mL) = 7245.2
Statistical Analysis 5: Comparison: Treatment C - 1000 mg Diabex; Geometric least squares means for Treatment C; Test type: Superiority or Other; Geometric Least Squares Mean (ng*hr/mL) = 11680
Statistical Analysis 6: Comparison: Treatment D - 1000 mg Glucophage; Geometric least squares means for Treatment D; Test type: Superiority or Other; Geometric Least Squares Mean (ng*hr/mL)] = 11641

2. Primary Outcome: Metformin PK Parameter Observed Maximum Plasma Concentration (Cmax)
Description: PK is the process by which a drug is absorbed, distributed, metabolized, and eliminated by the body. Cmax is the maximum observed concentration of drug substance in plasma.
Time Frame: Periods 1, 2, 3, & 4: pre-dosing, 15, 30, 45 mins & 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36 & 48 hrs post-dosing
Population: All treated participants with evaluable PK analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A - 500 mg Diabex | Treatment B - 500 mg Glucophage | Treatment C - 1000 mg Diabex | Treatment D - 1000 mg Glucophage
Number analyzed (Participants) | 28 | 27 | 27 | 26
ng/mL | 1013.57 (25.67) | 1019.59 (25.26) | 1635.30 (27.67) | 1593.20 (26.87)
Statistical Analysis 1: Comparison: Treatment A - 500 mg Diabex vs Treatment B - 500 mg Glucophage; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio (%) of Geometric LS Means = 101.12, 95% CI 2-sided [96.36 to 106.11] — Ratio=Treatment B/Treatment A. Geometric LS means values are presented in other statistical analysis entries
Statistical Analysis 2: Comparison: Treatment C - 1000 mg Diabex vs Treatment D - 1000 mg Glucophage; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio (%) of Geometric LS Means = 98.65, 95% CI 2-sided [93.94 to 103.59] — Ratio=Treatment B/Treatment A. Geometric LS means values are presented in other statistical analysis entries
Statistical Analysis 3: Comparison: Treatment A - 500 mg Diabex; Geometric least squares means for Treatment A; Test type: Superiority or Other; Geometric Least Squares Mean (ng/mL) = 1013.6
Statistical Analysis 4: Comparison: Treatment B - 500 mg Glucophage; Geometric least squares means for Treatment B; Test type: Superiority or Other; Geometric Least Squares Mean (ng/mL) = 1024.9
Statistical Analysis 5: Comparison: Treatment C - 1000 mg Diabex; Geometric least squares means for Treatment C; Test type: Superiority or Other; Geometric Least Squares Mean (ng/mL) = 1643.8
Statistical Analysis 6: Comparison: Treatment D - 1000 mg Glucophage; Geometric least squares means for Treatment D; Test type: Superiority or Other; Geometric Least Squares Mean (ng/mL) = 1621.6

3. Secondary Outcome: Participants With Adverse Events (AEs), Discontinuations Due to AEs, Deaths, and Serious AEs (SAEs)
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition in a subject administered an investigational product and that does not necessarily have a causal relationship with this treatment. SAE=any untoward medical occurrence that results in death, is life-threatening, requires or prolongs inpatient hospitalization (including elective surgery), results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event.
Time Frame: AEs: from study drug administration Day 1/Period 1 till study discharge. SAEs: from date of written consent until 30 days after discontinuation of dosing or study participation. Duration of the study was approximately 45 days (including screening).
Population: All treated participants not discontinuing prior to the end of the study.
Measure: Number; unit: Participants
Arm/Group | Treatment A - 500 mg Diabex | Treatment B - 500 mg Glucophage | Treatment C - 1000 mg Diabex | Treatment D - 1000 mg Glucophage
Number analyzed (Participants) | 28 | 27 | 27 | 27
Participants
  Participants With atleast 1 Treatment-emergent AE | 6 | 2 | 5 | 6
  Discontinuations Due to AE | 0 | 0 | 0 | 0
  Deaths | 0 | 0 | 0 | 0
  SAEs | 0 | 0 | 0 | 0

4. Secondary Outcome: Participants With Electrocardiogram Abnormalities Considered Clinically Significant or Reported as an AE
Description: Clinically significant was determined by the investigator. ECGs were recorded after participants had been supine for at least 5 minutes.
Time Frame: From study drug administration Day 1/Period 1 till study discharge. Duration of the study was approximately 45 days (including screening).
Population: All treated participants not discontinuing prior to the end of the study.
Measure: Number; unit: Participants
Arm/Group | Treatment A - 500 mg Diabex | Treatment B - 500 mg Glucophage | Treatment C - 1000 mg Diabex | Treatment D - 1000 mg Glucophage
Number analyzed (Participants) | 28 | 27 | 27 | 27
Participants | 0 (0) | 0 (0) | 0 (0) | 0 (0)

5. Secondary Outcome: Participants With Abnormal Physical Findings
Description: Physical findings that were considered abnormal by the investigator.
Time Frame: From Day 1/Period 1 to study discharge or premature discontinuation. Duration of study was approximately 45 days (including screening).
Population: All treated participants not discontinuing prior to the end of the study.
Measure: Number; unit: Participants
Arm/Group | Treatment A - 500 mg Diabex | Treatment B - 500 mg Glucophage | Treatment C - 1000 mg Diabex | Treatment D - 1000 mg Glucophage
Number analyzed (Participants) | 28 | 27 | 27 | 27
Participants | 0 | 0 | 0 | 0

6. Secondary Outcome: Participants With Abnormal Vital Sign Findings Reported as an AE
Description: per investigator
Time Frame: as for outcome 5
Population: All treated participants not discontinuing prior to the end of the study.
Measure: Number; unit: Participants
Arm/Group | Treatment A - 500 mg Diabex | Treatment B - 500 mg Glucophage | Treatment C - 1000 mg Diabex | Treatment D - 1000 mg Glucophage
Number analyzed (Participants) | 28 | 27 | 27 | 27
Participants | 0 | 0 | 0 | 0

7. Other Pre Specified Outcome: Metformin Pharmacokinetic (PK) Parameter Time to Achieve the Observed Maximum Plasma Concentration (Tmax)
Description: PK is the process by which a drug is absorbed, distributed, metabolized, and eliminated by the body. Tmax is the time taken to reach the maximum observed plasma concentration.
Time Frame: Periods 1, 2, 3, & 4: pre-dosing, 15, 30, 45 mins & 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36 & 48 hrs post-dosing
Population: All treated participants with evaluable PK analyses.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Treatment A - 500 mg Diabex | Treatment B - 500 mg Glucophage | Treatment C - 1000 mg Diabex | Treatment D - 1000 mg Glucophage
Number analyzed (Participants) | 28 | 27 | 27 | 26
hr | 3.25 (0.79) | 3.56 (0.80) | 3.22 (0.64) | 3.23 (0.80)

8. Other Pre Specified Outcome: Metformin Pharmacokinetic (PK) Parameter Terminal Half-life (T 1/2)
Description: PK is the process by which a drug is absorbed, distributed, metabolized, and eliminated by the body. T 1/2 is the time required for the concentration of the drug to reach half of its original value in plasma
Time Frame: Periods 1, 2, 3, & 4: pre-dosing, 15, 30, 45 mins & 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36 & 48 hrs post-dosing
Population: All treated participants with evaluable PK analyses. In treatment D, T 1/2 was not analysed for 1 participant who did not have a clear terminal elimination phase.
Measure: Mean (Standard Deviation); unit: hr
Groups:
- Treatment B - 500 mg Glucophage: Single oral dose of 500 mg Glucophage tablet administered in the fed condition
- Treatment C - 1000 mg Diabex: Single oral dose of 1000 mg Diabex tablet administered in the fed condition
- Treatment D - 1000 mg Glucophage: Single oral dose of 1000 mg Glucophage tablet administered in the fed condition
Arm/Group | Treatment A - 500 mg Diabex | Treatment B - 500 mg Glucophage | Treatment C - 1000 mg Diabex | Treatment D - 1000 mg Glucophage
Number analyzed (Participants) | 28 | 27 | 27 | 25
hr | 13.2310 (5.3180) | 11.5349 (3.7633) | 12.6152 (4.2032) | 12.5268 (4.3137)

9. Secondary Outcome: Participants With Clinical Laboratory Findings Considered Clinically Significant or Reported as an AE: Hematology
Description: Clinically significant was determined by the investigator.
Time Frame: as for outcome 4
Population: All treated participants not discontinuing prior to the end of the study.
Measure: Number; unit: Participants
Arm/Group | Treatment A - 500 mg Diabex | Treatment B - 500 mg Glucophage | Treatment C - 1000 mg Diabex | Treatment D - 1000 mg Glucophage
Number analyzed (Participants) | 28 | 27 | 27 | 27
Participants | 0 | 0 | 0 | 0

10. Secondary Outcome: Participants With Clinical Laboratory Findings Considered Clinically Significant or Reported as an AE: Serum Chemistry
Description: Clinically significant was determined by the investigator.
Time Frame: as for outcome 4
Population: All treated participants not discontinuing prior to the end of the study.
Measure: Number; unit: Participants
Arm/Group | Treatment A - 500 mg Diabex | Treatment B - 500 mg Glucophage | Treatment C - 1000 mg Diabex | Treatment D - 1000 mg Glucophage
Number analyzed (Participants) | 28 | 27 | 27 | 27
Participants | 0 | 0 | 0 | 0

11. Secondary Outcome: Participants With Clinical Laboratory Findings Considered Clinically Significant or Reported as an AE: Urinalysis
Description: Clinically significant was determined by the investigator.
Time Frame: as for outcome 4
Population: All treated participants not discontinuing prior to the end of the study.
Measure: Number; unit: Participants
Arm/Group | Treatment A - 500 mg Diabex | Treatment B - 500 mg Glucophage | Treatment C - 1000 mg Diabex | Treatment D - 1000 mg Glucophage
Number analyzed (Participants) | 28 | 27 | 27 | 27
Participants | 0 | 0 | 0 | 0

12. Other Pre Specified Outcome: Metformin Pharmacokinetic (PK) Parameter Area Under the Plasma Concentration Versus Time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUC[0-t])
Description: PK is the process by which a drug is absorbed, distributed, metabolized, and eliminated by the body. AUC[0-t] is the area under the plasma concentration-time curve from time zero to time of last measurable concentration.
Time Frame: Periods 1, 2, 3, & 4: pre-dosing, 15, 30, 45 mins & 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36 & 48 hrs post-dosing
Population: All treated participants with evaluable PK analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Treatment A - 500 mg Diabex | Treatment B - 500 mg Glucophage | Treatment C - 1000 mg Diabex | Treatment D - 1000 mg Glucophage
Number analyzed (Participants) | 28 | 27 | 27 | 26
ng*hr/mL | 6907.06 (27.16) | 7078.70 (26.18) | 11305.27 (27.77) | 11129.89 (28.93)
Statistical Analysis 1: Comparison: Treatment A - 500 mg Diabex vs Treatment B - 500 mg Glucophage; Test type: Superiority or Other; Ratio (%) of Geometric LS Means = 103.19, 95% CI 2-sided [99.75 to 106.75] — Ratio=Treatment B/Treatment A. Geometric LS means values are presented in other statistical analysis entries
Statistical Analysis 2: Comparison: Treatment C - 1000 mg Diabex vs Treatment D - 1000 mg Glucophage; Test type: Superiority or Other; Ratio (%) of Geometric LS Means = 99.44, 95% CI 2-sided [96.08 to 102.92] — Ratio=Treatment D/Treatment C. Geometric LS means values are presented in other statistical analysis entries
Statistical Analysis 3: Comparison: Treatment A - 500 mg Diabex; Geometric least squares means for Treatment A; Test type: Superiority or Other; Geometric Least Squares Mean (ng*hr/mL) = 6907.1
Statistical Analysis 4: Comparison: Treatment B - 500 mg Glucophage; Geometric least squares means for Treatment B; Test type: Superiority or Other; Geometric Least Squares Mean (ng*hr/mL) = 7127.4
Statistical Analysis 5: Comparison: Treatment C - 1000 mg Diabex; Geometric least squares means for Treatment C; Test type: Superiority or Other; Geometric Least Squares Mean (ng*hr/mL) = 11391
Statistical Analysis 6: Comparison: Treatment D - 1000 mg Glucophage; Geometric least squares means for Treatment D; Test type: Superiority or Other; [Geometric Least Squares Mean (ng*hr/mL) = 11327

ADVERSE EVENTS:
Time Frame: From study drug administration Day 1/Period 1 till study discharge. Duration of the study was approximately 45 days (including screening).
Arm/Group | Treatment C - 1000 mg Diabex | Treatment D - 1000 mg Glucophage | Treatment A - 500 mg Diabex | Treatment B - 500 mg Glucophage
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/28 | 0/27
Other Adverse Events (participants affected / at risk) | 5/27 | 6/27 | 6/28 | 2/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment C - 1000 mg Diabex (N=27) | Treatment D - 1000 mg Glucophage (N=27) | Treatment A - 500 mg Diabex (N=28) | Treatment B - 500 mg Glucophage (N=27)
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 2 | 4 | 2 | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Feeling of body temperature change (General disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication